CLINICAL TRIAL: NCT01592188
Title: Cognitively-Based Compassion Training and Mindfulness Attention Training for Elementary School Students
Brief Title: Cognitively-Based Compassion Training and Mindfulness Attention Training Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thaddeus Pace, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IRB00054782; CBCT-Paideia (Other: Other)
Record Dates: First submitted 2012-05-02; First posted 2012-05-07 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Behavioral Resilience; Biological Resilience
Keywords: meditation, inflammation, children, attention
MeSH Terms: conditions — Inflammation | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MT (Active Comparator): Mindfulness training. Participants will be provided with once per week training in mindfulness meditation.
  Interventions: Behavioral: Mindfulness training
- CBCT (Experimental): Cognitively-based compassion training. Participants in this arm will be provided with once weekly training on the cognitively-based compassion training program.
  Interventions: Behavioral: Cognitively-Based Compassion Training (CBCT)

INTERVENTIONS:
Behavioral: Cognitively-Based Compassion Training (CBCT) — CBCT is a 12 week program that begins by teaching mindfulness and attention. It then goes on to use new mindfulness skills to consider topics of compassion, or unbiased acceptance and compassion for all other people, both friends, unfamiliar people, and enemies.
  Other Names: Compassion Meditation
  Arms: CBCT
Behavioral: Mindfulness training — Mindfulness training will consist of 6 weeks training in mindfulness meditation.
  Other Names: Mindfulness meditation
  Arms: MT

SUMMARY:
This project will explore the effect of Cognitively-Based Compassion Training or mindfulness training on behavior and saliva stress hormones in elementary school-age children.

DETAILED DESCRIPTION:
This project will explore the effect of Cognitively-Based Compassion Training (CBCT) or mindfulness training (MT) on different aspects of behavior and stress-related biology in elementary school-age children. The program will consist of 12 weeks of CBCT or MT, and various social behavioral assessments will be conducted. Participants will also provide saliva in which concentrations of stress hormones including cortisol and the inflammatory biomarkers C-reactive protein will be measured.

ELIGIBILITY:
Inclusion Criteria:

* age 7-12
* enrollment at the Paideia School.

Exclusion Criteria:

* poor physical health
* enrollment at a school other than the Paideia school.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Interpersonal behaviors assessed using standardized protocols of social behavior, social cognition, and empathy. | 12 weeks
  Assessments before and after CBCT or MT interventions will be conducted to see if these practices lead to changes in interpersonal behavior. Participants will be asked to respond to questions related to social behavior in the lab setting, with the Social Circle Task, Mind In The Eyes Task, and the Implicit Association Task.
Concentrations of stress system biomarkers in saliva | 12 weeks
  Assessments before and after CBCT or MT interventions will be conducted to see if these practices lead to changes in stress system activity, as measured by key biomarkers (cortisol, C-reactive protein) in saliva samples.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rochat, PhD, Principal Investigator — Emory University; Thaddeus Pace, PhD, Principal Investigator — Emory University
Locations (1):
- Paideia School, Atlanta, Georgia, United States